CLINICAL TRIAL: NCT00004788
Title: Study of Nutritional Factors in Porphyria
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11886; UTMB-328
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Porphyria
Keywords: inborn errors of metabolism; porphyria; rare disease
MeSH Terms: conditions — Porphyrias; Metabolism, Inborn Errors; Rare Diseases

SUMMARY:
OBJECTIVES: I. Determine whether differences in dietary habits are associated with disease activity in patients with acute intermittent porphyria.

II. Determine whether premenstrual porphyria attacks are associated with increased luteal phase energy requirements.

III. Determine whether energy requirements are higher than intakes in men with unexplained frequent porphyria attacks.

IV. Assess the nutritional status of women with acute intermittent porphyria using a comprehensive series of laboratory methods, including zinc and pyridoxine status.

V. Determine whether the frequency of disease exacerbations decreases when dietary and nutritional abnormalities are corrected in these patients.

VI. Evaluate the safety and efficacy of a parenteral nutrition regimen for patients with acute porphyria attacks.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Women record diet intake for at least 1 cycle (28 days), then undergo a comprehensive nutritional assessment at least once during the follicular and luteal phases of the cycle.

Men also record diet intake for at least 1 month and undergo indirect calorimetry and other studies.

All patients receive a comprehensive analysis of diet and energy metabolism. Energy expenditure, resting metabolic rates, and basal metabolic rates are determined with indirect calorimetry, including measurements taken during the follicular and luteal phases of the cycle. Other testing includes hormone assays, serology for nutritional studies, and a urinary metabolite profile. Zinc, lead, and other metals are measured by atomic absorption spectroscopy.

The diagnosis of acute intermittent porphyria is confirmed by erythrocyte porphobilinogen deaminase; urinary aminolevulinic acid, porphobilinogen, and porphyrins; and total fecal porphyrins.

Patients hospitalized for acute attacks of porphyria during the study will receive standard treatment, including intravenous hematin and parenteral support.

ELIGIBILITY:
* Acute intermittent porphyria
* Variegate porphyria and hereditary coproporphyria eligible but analyzed separately

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1988-05

CONTACTS AND LOCATIONS:
Overall Officials: Karl Elmo Anderson, Study Chair — University of Texas